CLINICAL TRIAL: NCT02263989
Title: Bioequivalence of the 40 mg Telmisartan Film-coated Tablet Compared With the Conventional 40 mg Telmisartan Tablet Following Oral Administration in Healthy Male Volunteers (an Open-label, Randomised, Single-dose, Two-sequence, Four-period Replicated Crossover Study)
Brief Title: Bioequivalence of Telmisartan Film-coated Tablet Compared With the Conventional Telmisartan Tablet Following Oral Administration in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 502.520
Record Dates: First submitted 2014-10-13; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan

ARMS (2):
- Telmisartan film coated tablet (Experimental)
  Interventions: Drug: Telmisartan film coated tablet
- Telmisartan conventional tablet (Active Comparator)
  Interventions: Drug: Telmisartan conventional tablet

INTERVENTIONS:
Drug: Telmisartan film coated tablet
  Arms: Telmisartan film coated tablet
Drug: Telmisartan conventional tablet
  Arms: Telmisartan conventional tablet

SUMMARY:
Study to investigate the bioequivalence of the 40 mg telmisartan film-coated tablet vs. the conventional 40 mg telmisartan tablet

ELIGIBILITY:
Inclusion Criteria:

Healthy males according to the following criteria:

1. Based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate, body temperature), 12-lead ECG, clinical laboratory tests

   * No findings deviating from normal and of clinical relevance
   * No evidence of a clinically relevant concomitant disease
2. Age ≥20 and ≤35 years
3. Body mass index (BMI) ≥17.6 and ≤26.4 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
3. Chronic or relevant acute infections
4. Any clinical relevant findings of the laboratory test deviating from normal
5. Positive result for either hepatitis B surface antigen (HBs antigen), anti hepatitis C virus (HCV) antibodies, syphilitic test or human immunodeficiency virus (HIV) test
6. History of surgery of gastrointestinal tract (except appendectomy)
7. History of relevant orthostatic hypotension (mean standing systolic blood pressure (SBP) varies by ≥20 mmHg from mean supine SBP or mean standing diastolic blood pressure (DBP) varies by ≥10 mmHg from mean supine DBP), fainting spells or blackouts
8. History of hepatic dysfunction (e.g. biliary cirrhosis, cholestasis)
9. History of serious renal dysfunction
10. History of bilateral renal artery stenosis or renal artery stenosis in a solitary kidney
11. History of cerebrovascular disorder
12. History of hyperkalemia
13. Known hypersensitivity to any component of the telmisartan formulation, or to any other angiotensin II receptor blockers (ARBs)
14. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
15. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 7 days prior to administration or during the trial
16. Participation in another trial with an investigational drug within 4 months or 6 half-lives of the investigational drug prior to administration
17. Smoker (≥20 cigarettes/day)
18. Alcohol abuse (60 g or more ethanol/day: ex. 3 middle-sized bottles of beer, 3 gous (equivalent to 540 mL) of sake)
19. Drug abuse
20. Blood donation (more than 100 mL within 4 weeks prior to administration or during the trial)
21. Excessive physical activities (within 1 week prior to administration or during the trial)
22. Intake of alcohol within 2 days prior to administration
23. Inability to comply with dietary regimen of study centre
24. Inability to refrain from smoking on trial days

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to last quantifiable data point) | up to 72 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours after drug administration

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours after drug administration
tmax (time from dosing to the maximum measured concentration of the analyte in plasma) | up to 72 hours after drug administration
λz (terminal rate constant of the analyte in plasma) | up to 72 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 72 hours after drug administration
MRTpo (mean residence time of the analyte in the body after po administration) | up to 72 hours after drug administration
Number of subjects with adverse events | up to 72 hours after last administration
Number of subjects with clinically significant findings in vital signs | up to 72 hours after last administration
  blood pressure, pulse rate, body temperature
Number of subjects with clinically significant findings in 12-lead electrocardiogram | up to 72 hours after last administration
Number of subjects with clinically significant findings in laboratory tests | up to 72 hours after last administration
Number of subjects with clinically significant findings in physical examination | up to 72 hours after last administration